CLINICAL TRIAL: NCT00333515
Title: A Phase 1, Randomized, Observer-blinded, Single Dose, Placebo Controlled Dosage-Escalation Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Plasma-Derived Human Butyrylcholinesterase (HuBChE) Administered Intravenously (IV)
Brief Title: Pharmacokinetic (PK) and Safety Study of Plasma-derived Human Butyrylcholinesterase Administered Intravenously
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Collaborators: DynPort Vaccine Company LLC, A GDIT Company (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: HuBChE-01
Record Dates: First submitted 2006-06-01; First posted 2006-06-05 (Estimated); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Healthy Volunteers; Chemical Terrorism; Chemical Warfare
Keywords: Chemical nerve agent intoxication

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Administration of one of 3 doses (dose escalation) of the active drug (HuBChE). (Dose-escalation proceeds only after safety evaluation and after the previous dosage has been found to be acceptable by an independent Data Safety Monitoring Board.)
  Interventions: Drug: Human Butyrylcholinesterase (HuBChE) derived from human plasma
- 2 (Placebo Comparator): Administration of placebo
  Interventions: Drug: Placebo: Normal saline

INTERVENTIONS:
Drug: Human Butyrylcholinesterase (HuBChE) derived from human plasma — Administration via IV infusion at a rate of 50 mg/min (2 mL/min)
  Arms: 1
Drug: Placebo: Normal saline — Administration via IV infusion at a rate of 50 mg/min (2 mL/min)
  Arms: 2

SUMMARY:
The purpose of this placebo-controlled study is to evaluate the safety, tolerability and pharmacokinetics of a single dose regimen of human butyrylcholinesterase (HuBChE) in healthy adults at 3 ascending dosage levels administered IV. HuBChE, which occurs naturally in human plasma, is being evaluated for prophylaxis and treatment in the event of exposure to chemical nerve agents (as employed during chemical warfare or as an act of terrorism). Volunteers in each dosage cohort will be randomized to treatment with HuBChE active drug or normal saline placebo in a 3:1 ratio. The volunteers will remain in the study for 90 (+/- 7) days. For the first 3 days following dose administration, they will remain at the clinical trial site as inpatients and will be closely monitored for patient safety. Afterwards, they will return to the trial site (at pre-determined intervals) as outpatients for 8 further visits, where patient safety will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* The volunteer is between 18 and 55 years of age (inclusive) at the time of administration of HuBChE.
* The volunteer is in good health as determined by the Investigator (Study Doctor) from a medical history and physical examination.
* The volunteer has clinical chemistry, hematology, coagulation, and urinalysis laboratory values within acceptable ranges or deemed clinically insignificant by the Principal Investigator (PI) and Project Medical Monitor.
* The volunteer has a normal electrocardiogram (ECG) or one with clinically insignificant findings as deemed by the PI.
* The volunteer is willing to have his or her blood samples stored for future HuBChE research studies.
* The volunteer has signed the Informed Consent form (ICF) and has signed the Health Insurance Portability and Accountability Act (HIPAA) authorization form.
* The volunteer agrees not to donate blood during the trial or for at least 2 months following the 90 day study visit.
* The volunteer is willing to comply with the requirements of the protocol through the post-infusion Day 90 (± 7 days) visit.
* Female volunteers must be of non-childbearing potential (i.e., surgically sterilized or postmenopausal), or must not be pregnant (as indicated by a negative urine pregnancy test within 1 day prior to HuBChE administration) or nursing, and must use two types of acceptable forms of Food and Drug Administration (FDA)-approved birth control methods, including:

  * Progesterone only hormonal types of birth control (such as implants or birth control pills) or an intrauterine device (IUD) and
  * an additional barrier type of birth control measure (i.e., condoms, diaphragms, cervical caps, etc.) during the period beginning from 30 days before HuBChE administration through completion of the study. Completion of the study is defined as completing the acute phase of the study (Day 45 [± 3 days] visit).

Exclusion Criteria:

* The volunteer demonstrates predisposition to thrombus formation as determined by past medical history, and family history.
* The volunteer has a history of anaphylactoid reaction or other serious adverse reactions to blood products.
* The volunteer has a history of allergic reaction to procainamide or to its metabolite, p-aminobenzoic acid.
* The volunteer has been diagnosed with alcohol or drug abuse within the 12 months prior to study screening or offers a history of alcohol or drug abuse within the 12 months prior to screening.
* The volunteer has a positive result on a urine drug screen that tests for common substances of abuse, such as amphetamines, barbiturates, benzodiazepines, cocaine, opiates, and cannabinoids. (If positive on screen, confirmatory testing shall be performed where applicable.)
* The volunteer has a previous diagnosis of any serious psychiatric disorder. For this purpose, serious psychiatric disorder is defined as illness requiring hospitalization within the previous 12 months; routine administration of more than one medication to control anxiety, mood or sleep disorder; or history of suicide attempt.
* The volunteer has received any blood products or immune globulin in the previous six months.
* The volunteer has donated blood within 56 days prior to receipt of study product (Day 0).
* The volunteer has a deficiency of immunoglobulin A (IgA) as determined on screening.
* The volunteer has a current or past medical history for any condition which, in the opinion of the PI and/or Project Medical Monitor (PMM), might place him or her at risk by participating in the study.
* Personal or family history (in first degree relatives) of significant neuromuscular disease (as determined by the PI).
* Female volunteer is pregnant (must have a negative urine pregnancy test within 1 day of receipt of HuBChE), lactating, or unwilling to use 2 types of an acceptable FDA-approved form of contraception from time of screening through completion of the Day 45 (± 1 day) study visit.
* Current use, receipt within the previous 14 days, or intent to use during the 14 days after receiving drug product of drugs that may be metabolized, inhibited, or otherwise affected by BChE.
* The volunteer has a clinically significant abnormality on the ECG.
* The volunteer has any laboratory values outside acceptable ranges that are clinically significant as assessed by the Investigator and/or PMM. The volunteer tests positive for HIV, HCV, or HBV at screening.
* The volunteer has an acute illness, evidence of significant active infection, or evidence of systemic disease at time of enrollment that in the opinion of the PI would place the volunteer at an unacceptable risk for injury.
* The volunteer has a temperature >100.4°F at the time of dose administration.
* The volunteer has occupational or other responsibilities that would prevent completion of participation in the study.
* The volunteer is currently using tobacco products.
* Participants in other clinical trails in the past 60 days.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2008-04-01 (Actual); Study Completion 2008-08-01 (Actual)

PRIMARY OUTCOMES:
Frequence and severity of local and systemic AEs | until post-infusion Day 90 (+/- 7 days)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Quintiles Phase 1 Services, Lenexa, Kansas, United States